CLINICAL TRIAL: NCT06752330
Title: Evaluation of the Effect of a Probiotic in Subjects Undergoing Fixed Orthodontic Appliances With Multibrackets or Clear Aligners: a Single-blind Randomized Controlled Trial
Brief Title: Evaluation of the Effect of a Probiotic in Patients Undergoing Orthodontic Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Turin, Italy (Other)
Responsible Party: Principal Investigator, Jacopo Lanzetti, Dental Hygienist, University of Turin, Italy
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 0001105
Record Dates: First submitted 2024-12-20; First posted 2024-12-30 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Orthodontics; Dental Hygiene; Gingivitis and Periodontal Diseases
Keywords: probiotics; Fixed orthodontic; oral hygiene; clear aligners
MeSH Terms: conditions — Gingivitis; Periodontal Diseases

STUDY DESIGN:
Who Masked: Investigator
Masking Description: The operator performing the data collection was unaware of the group membership of the evaluated patient
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Domiciliary oral hygiene with probiotics (Experimental): During the first sitting (T0), after checking the inclusion criteria to enter the re-search protocol, a professional oral hygiene session is carried out through the use of ultrasonic inserts, hand instruments, and glycine powder.
  One month after the first session (T1), FMPS and FMBS are detected. Probiotic administration is discontinued in patients belonging to the test group.
  At 2 months from baseline (T2), plaque and bleeding indices are recalculated and, for test group patients only, probiotic supply is delivered for 1 month.
  Then, after 1 month (T3), plaque and bleeding indices are measured and probiotic supply is discontinued.
  Interventions: Dietary Supplement: Use of probiotics during oral hygiene at home
- Domiciliary oral hygiene alone (No Intervention): During the first sitting (T0), after checking the inclusion criteria to enter the re-search protocol, a professional oral hygiene session is carried out through the use of ultrasonic inserts, hand instruments, and glycine powder. All patient is instructed to perform home oral hygiene procedures using a medium-bristle manual toothbrush and fluoride toothpaste (1450 ppm F) with no added anti-plaque or anti-calculus property. Patients are advised against the use of any mouthwash.

INTERVENTIONS:
Dietary Supplement: Use of probiotics during oral hygiene at home — The probiotic used in the study is Bifidobacterium Lactis HN019, distributed com-mercially in Italy by Curasept (Curasept Prevent®, Curasept S.p.A., Saronno, VA, Italy), with added Kluyveromyces Marxianus Fragilis B0399, colostrum and biotin. The probiotic was taken by patients following the manufacturer's directions via 2 chewable tablets daily, morning and evening, after normal daily oral hygiene, achieving daily average values of B. Lactis HN019 of 2*107 CFU and Kluyveromyces marxianus fragilis B0399 of 2*109 CFU.
  Arms: Domiciliary oral hygiene with probiotics

SUMMARY:
Orthodontic patients need supplementary oral hygiene tools in addition to professional oral hygiene. The aim of this study is to evaluate the effects of Bifidobacterium animalis subs. Lactis HN019 on plaque accumulation and gingival bleeding in orthodontic patients.

ELIGIBILITY:
Inclusion Criteria:

* age range of 10 to 30 years old;
* good general health;
* patients undergoing fixed multibracket orthodontic treatment;
* patients undergoing invisible aligner orthodontic treatment.

Exclusion Criteria:

* physical, mental or motor disabilities;
* systemic conditions that influence the progression of gingivitis;
* presence of non-plaque-induced gingivitis;
* known allergies;
* smokers (if more than 5 cigarettes per day);
* use of antibiotics, anti-inflammatories, or probiotics in the 6 months prior to recruitment.

Ages: 10 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Actual)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Full Mouth Bleeding Score (FMBS) | 4 months
  FMBS is a dichotomous index indicating the presence of gingival bleeding on 6 surfaces, the same as FMPS, after light probing. The ratio of surfaces with bleeding to the total of the assessed surfaces is presented as a percentage.

SECONDARY OUTCOMES:
Full Mouth Plaque Score (FMPS) | 4 months
  FMPS is a dichotomous index indicating the presence of bacterial biofilm on 6 tooth surfaces: mesio-vestibular, vestibular, disto-vestibular, disto-palatal/lingual, pala-tal/lingual, and mesio-palatal/lingual. The ratio of surfaces with plaque to the total of the assessed surfaces is presented as a percentage.

CONTACTS AND LOCATIONS:
Locations (1):
- AOU Città della Salute e della Scienza, Torino, Italy, Italy

IPD SHARING:
Plan to Share IPD: Yes
IPD will shared by papers or presentations
Supporting Information: Study Protocol, SAP, ICF, CSR